CLINICAL TRIAL: NCT07162779
Title: Evaluation of [68Ga]DOTA-IR-780-C-4 in PET Imaging Studies for PSMA-Positive Prostate Cancer Patients
Acronym: PSMA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2025002; 22274074 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-07-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: PET CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET imaging of primary and metastatic lesions in prostate cancer patients (Experimental): [68Ga]DOTA-IR-780-C-4 is administered through a superficial vein on the back of the hand. A PET/CT scan was performed approximately 1 h, 2 h and 3 h after injection
  Interventions: Drug: Radioactive drugs are administered through intravenous injection.

INTERVENTIONS:
Drug: Radioactive drugs are administered through intravenous injection. — [68Ga]DOTA-IR-780-C-4 is administered through a superficial vein on the back of the hand. A PET/CT scan was performed approximately 1 h,2 h and 3 h after injection

SUMMARY:
Prostate cancer is one of the most common malignant tumors in the urinary and male reproductive systems. According to the 2020 edition of the Global Cancer Statistics Report published by the WHO International Agency for Research on Cancer in February 2021, newly diagnosed prostate cancer cases worldwide accounted for 7.3% of all malignant tumors in 2020, with an incidence rate ranking third after breast cancer and lung cancer. Deaths from prostate cancer accounted for 3.8% of all malignant tumor deaths, ranking eighth. In January 2019, the National Cancer Center released the latest incidence and mortality data of malignant tumors in China in 2015. Among them, there were 72,000 new prostate cancer cases, with an incidence rate of 10.23 per 100,000, ranking sixth among male malignant tumors; 31,000 deaths, with a mortality rate of 4.36 per 100,000, ranking tenth among male malignant tumors. Compared with European and American countries, prostate cancer in China has a relatively high mortality rate, mainly because most patients are diagnosed at an advanced stage. "Early diagnosis and early treatment" are important means to prolong the survival period and reduce the mortality rate of prostate cancer patients. Currently, the diagnostic methods for prostate cancer mainly include digital rectal examination, tumor markers, imaging examinations, and prostate biopsy.

Prostate-specific membrane antigen (PSMA) is a type II transmembrane glycoprotein secreted by prostate epithelial cells, which is highly expressed in the cell membrane of prostate cancer cells and their metastases. PSMA is also weakly expressed in normal tissues such as the small intestine, brain, kidneys (proximal convoluted tubules), duodenal mucosa, parotid gland, and submandibular gland, but only at 1/1000 to 1/100 of the level in prostate cancer. Bostwick et al. used the PSMA-targeting antibody 7E11-C5 to detect tissues from 184 patients with prostate cancer lesions and found that the staining intensity was higher in prostate cancer tissues with higher Gleason scores. Subsequent studies by Silver et al. also found that the expression level of PSMA in prostate cancer tissues is much higher than that in normal prostate tissues, and its expression level is significantly correlated with the pathological stage of prostate cancer, with an expression rate of up to 96%-98% in lymph node metastases. The specific high expression of PSMA in cancer tissues makes it an important target for the diagnosis and treatment of prostate cancer, and a large number of radioactive molecular probes have been developed targeting this target for the diagnosis of prostate cancer, showing good target affinity.

The properties of different PSMA radiotracers vary slightly. Inhibitors of PSMA are mainly divided into three categories: phosphorous-based, thiol-based, and urea-based. Among them, the most widely used PSMA PET imaging agents are urea-based small molecules, such as 68Ga-PSMA-11, 68Ga-PSMA-617, 68Ga-PSMA-I&T, 18F-DCFBC, 18F-DCFPyL, and 18F-PSMA-1007. Multiple studies have shown that compared with other PET imaging modalities or traditional imaging, PSMA PET imaging has significant advantages, including higher specificity, sensitivity, and positive predictive value.

68Ga-labeled PSMA ligands, as the first PSMA PET imaging agents applied to prostate cancer, have shown promising prospects in tumor localization, local staging, detection of biochemical recurrence (BCR), metastasis detection, and guiding treatment. Among these ligands, PSMA-11 is the most clinically used. 68Ga-PSMA-11 was approved by the FDA in December 2020. It is very helpful for prostate cancer patients with suspected metastasis or recurrence. For suspected metastases and recurrence, it can specifically bind to PSMA, clearly visualize lesions in PET imaging, accurately detect potential foci, provide important diagnostic basis for clinical practice, and assist doctors in judging disease progression and formulating effective treatment plans.

Another similar product, Pluvicto, was approved by the FDA in March 2022. It is used for patients with suspected metastatic prostate cancer scheduled for initial radical treatment, patients with suspected recurrent prostate cancer with elevated PSA levels, and screening metastatic prostate cancer patients eligible for 177Lu-PSMA-617 targeted therapy.

In summary, this product shares the same target and nuclide (68Ga) as Pluvicto, and is expected to have obvious diagnostic performance in PSMA-positive prostate cancer. The experimental results of Pluvicto have demonstrated acceptable safety and good effectiveness of the drug, thus ensuring the safety and effectiveness of this probe.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the written Informed Consent Form (ICF); Willing and able to participate in procedures required by the trial, including examinations and follow-ups; Male, aged ≥ 18 years;

Histologically or cytologically confirmed prostate cancer, with failure of standard treatment, refusal of standard treatment, no available standard treatment, or disease progression after refractory previous treatments, or no available treatment options according to current guidelines:

Patients who have not received, refused to receive, or progressed after receiving at least 1 but no more than 2 taxane-based treatments. The taxane treatment regimen must include exposure to taxanes for at least 2 cycles. If the subject has only received one type of taxane and the doctor deems that he is not suitable for a second taxane treatment regimen (e.g., due to assessment of old age or health status indicating non-frailty or intolerance, etc.), he may also be included; Patients who have progressed after receiving at least one novel androgen-targeted drug (such as abiraterone, enzalutamide);

Meet the Prostate Cancer Working Group 3 (PCWG3) criteria for diagnosis of metastatic castration-resistant prostate cancer (mCRPC), including:

1. Serum testosterone reaches castration level (serum testosterone < 50 ng/dL or 1.7 nmol/L);
2. And at least one of the following:

Serum PSA progression: PSA > 1 ng/mL, and PSA increases consecutively twice at 1-week intervals, with both values exceeding 50% of the lowest value; or bone scan indicates ≥ 2 new bone lesions; or CT or MRI indicates progression of soft tissue lesions (RECIST 1.1) Confirmed as PSMA-positive by 68Ga-PSMA PET/CT scan; At least one measurable lesion (RECIST 1.1); Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2; Expected survival > 6 months;

Sufficient organ function:

1. Bone marrow function: neutrophil count ≥ 1.5 × 109/L; white blood cell count ≥ 2.5 × 109/L; platelet count ≥ 100 × 109/L; hemoglobin ≥ 90 g/L;
2. Liver function: total bilirubin ≤ 1.5 × ULN; albumin ≥ 30 g/L; ALT and AST < 3 × ULN in subjects without liver metastasis; < 5 × ULN in those with liver metastasis;
3. Renal function: creatinine clearance ≥ 60 mL/min calculated by the Cockcroft-Gault formula;
4. Coagulation function: INR ≤ 1.5; activated partial thromboplastin time (APTT) ≤ 2 × ULN (for patients not receiving anticoagulant therapy or receiving stable-dose anticoagulants); All clinically significant toxic reactions related to previous anti-tumor treatments (such as chemotherapy, radiotherapy, etc.) have recovered to ≤ Grade 1 (CTCAE V5.0) (except alopecia).

Agree to take radiation protection measures as directed by the doctor during the trial.

Exclusion Criteria:

Unable to tolerate imaging procedures; Having received other investigational drugs or devices within 4 weeks prior to screening; Having received any of the following treatments within 6 months prior to administration: radium-223, strontium-89, samarium-153, rhenium-188, or hemibody radiotherapy; Having previously received PSMA-targeted radioligand therapy; or having received systemic anticancer therapy such as radiotherapy, chemotherapy, immunotherapy, or biotherapy within 4 weeks prior to the first administration; Having experienced grade 4 myelosuppression after previous anticancer treatment, or grade 3 myelosuppression that required more than 6 weeks to recover; Planning to use cytotoxic chemotherapeutic drugs, antitumor immunotherapy, radioligand therapy, or other similar antitumor drugs during the trial; Having used blood products, albumin, etc. within half a month prior to administration to make the subject meet the inclusion criteria;

Having brain metastases, meningiomas, or other central nervous system metastases at screening, except for the following cases:

For asymptomatic brain metastases, where the metastatic lesions are limited to the supratentorial and/or cerebellum (i.e., no metastases in the midbrain, pons, medulla oblongata, or spinal cord), no corticosteroid treatment is needed, and there are no brain metastases with a long diameter > 1.5 cm, the subject can participate in the study; For symptomatic brain metastases, those who have received treatment and whose lesions are confirmed to be stable for more than 4 weeks by imaging can participate in the study; Having other malignant tumors within 5 years (except for locally treated malignant tumors in situ, such as basal cell or squamous cell skin cancer); Having superscan; Having symptomatic spinal cord compression or expected to develop spinal cord compression; Having previously received external beam radiation therapy (EBRT) targeting extensive bone marrow (>25%); Having undergone allogeneic organ transplantation and requiring immunosuppressive therapy;

Having severe heart disease at screening, including but not limited to the following:

QTcF > 470 ms or a history of long QTc; Having myocardial infarction, angina pectoris, coronary artery bypass grafting, etc. within 6 months prior to screening, which the investigator deems unsuitable for inclusion; Having any other diseases, metabolic abnormalities, physical examination abnormalities, or laboratory test abnormalities at screening, which, in the investigator's judgment, reasonably suggest a disease or state unsuitable for the use of the study drug, may affect the interpretation of study results, or put the subject at high risk; Having poorly controlled bladder outlet obstruction or urinary incontinence at screening; Having positive hepatitis C virus antigen (HCVAg) or human immunodeficiency virus antibody (HIV) at screening; For those with positive hepatitis B surface antigen (HBsAg) at screening, hepatitis B virus deoxyribonucleic acid (HBV-DNA) testing is required; if the investigator determines that the patient is in the active viral replication stage, they cannot be included; Having active infection prior to administration; Having poor venous conditions at screening and unable to tolerate blood sample collection; Having known allergies to protein and/or polypeptide drugs, or to structural analogs of this product or other excipients; Having a history of drug or alcohol abuse within one year prior to screening, or a long-term history of drug addiction; Failing to take effective contraceptive measures during sexual activity during the trial and within 6 months after the last administration.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
The dection performance of radiotracer [68Ga]DOTA-IR-780-C-4 | 1-2 hours
  precise PET imaging and diagnosis of primary and metastatic lesions in prostate cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangnan University Affiliated Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Protecting patient privacy

REFERENCES:
- See also: Related Info — https://www.medicalresearch.org.cn/login